CLINICAL TRIAL: NCT06791317
Title: Does Checklist Utilisation Decrease Complications Related to Intubation of the Critically Ill Adult? - a Two-phase Retrospective Study
Brief Title: Intubation Checklist in the Intensive Care Unit
Acronym: CHECC
Status: Active, not recruiting | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Jessica Kåhlin, Research group leader, Karolinska University Hospital
Other Study IDs: K2023-5312
Record Dates: First submitted 2025-01-15; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Critical Illness; Respiratory Failure; Unconsciousness
MeSH Terms: conditions — Critical Illness; Respiratory Insufficiency; Unconsciousness | interventions — Checklist

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard care: Intubation procedure before introduction of a checklist
  Interventions: Other: Checklist
- Checklist group: Intubation procedure after introduction of a checklist
  Interventions: Other: Checklist

INTERVENTIONS:
Other: Checklist — A checklist for the intubation procedure was organised into the categories physiological optimisation, equipment and drugs, team line-up, and contingency plan. This checklist was implemented in the clinic.

SUMMARY:
This retrospective study aims to explore whether the introduction of a preprocedural checklist for intubation in the intensive care unit (ICU) is associated with a lower incidence of intubation-related complications. Using a database where protocols from intubations in the ICU before implementing a checklist and after we will investigate whether a checklist affects early desaturation and hypotension after intubation.

DETAILED DESCRIPTION:
PROJECT PLAN

Does checklist utilisation decrease complications related to intubation of the critically ill adult? - a two-phase study

Study code: CHECC (Checklist for Endotracheal intubation in the Critical Care)

Ethical approval: This study will be conducted in accordance with GCP and National Swedish standards, as well as local standard procedures at the Clinical Research Unit at Function Perioperative Medicine and Intensive Care, Karolinska University Hospital and Karolinska Institutet, Stockholm, Sweden.

Principal investigator: Jessica Kåhlin, MD, PhD

Investigators:

Atosa Nejatian, MD Ida-Maria Forsberg, MD, PhD Malin Jonsson Fagerlund, MD, Assoc Professor

Affiliations for the above:

Perioperative Medicine and Intensive Care (PMI), Karolinska University Hospital and Department of Physiology and Pharmacology, Section for Anesthesiology and Intensive Care Medicine, Karolinska Institutet, Stockholm, Sweden

Background Endotracheal intubation is one of the most frequently performed procedures in the intensive care setting. However, it is associated with an alarmingly high incidence of complications. A recent study of emergency intubations performed in the intensive care unit (ICU), emergency department and wards found that approximately 40% resulted in intubation-related major adverse events, more commonly hypotension and hypoxemia. In addition, cardiac arrest was seen in 3% of intubations. These findings suggest that although endotracheal intubation is a common procedure, it still present a significant hazardous risk for the patient.

Preprocedural checklists have been used and implemented in various aspects and settings of health care. Among others, implementing a surgical checklist resulted in lower morbidity and mortality and in the ICU, using a checklist in conjunction with the placement of a central venous line significantly reduced central line-associated bloodstream infections.

A study on implementing a preprocedural intubation checklist on trauma patients in the emergency department showed a reduction in intubation-related complications such as oxygen desaturation, hypotension.

Checklists are a cognitive aid and practical tool to help planning and optimising a procedure systematically and set order. They promote standardisation and reduce reliance on individual memory, which can be compromised by stress and fatigue. This is used in aviation, product management and different healthcare areas. It usually contains a list of required items or suggestions and serves as a reminder how to optimise the patient, preferably with a contingency plan. Hence, in theory, this makes endotracheal intubation an ideal procedure for applying the checklist in critical ill patients in the ICU.

Intubation of the critically ill adult is associated with a significant risk of major complications, with patients having a limited physiological reserve, presenting a unique challenge for the intensivist. Guidelines advocate the employment of structured checklists for intubation. Preprocedural checklists have been used and significantly improved patient care in other aspects of health care. However, the number of studies on intubation checklists in the intensive care setting is currently limited, with contradictory results.

Therefore, we aim to investigate whether implementing a preprocedural intubation checklist in the ICU reduces in intubation-related complications in critically ill adults.

Objectives and purpose

This study aims to explore whether the introduction of a preprocedural checklist for intubation in the intensive care unit is associated with a lower incidence of intubation-related complications. The researchers hypothesise that the introduction and utilisation of a checklist will contribute to a safer and more structured working climate, leading to an optimised surrounding environment and enhanced physiology of the patient.

Research question

The primary hypothesis is that implementing a checklist for intubation in the intensive care will reduce hypoxemic and hypotensive events. The secondary hypothesis is that a checklist will reduce other adverse events, such as severe arrhythmias or fatal outcomes.

Primary endpoint:

Intubation-related complications:

* Peripheral oxygen saturation (SpO2) below 90% (or >5% drop if saturation is <90% after preoxygenation).
* Hypotension with systolic arterial blood pressure below 90 mmHg.

Secondary endpoints:

Does the implementation of a checklist for intubation result in the following:

* Decreased: 30-day mortality, ventilator days, ventilator-associated pneumonia, days in the ICU?
* A decreased number of intubation attempts and a higher first-pass success rate?
* A higher lowest median SpO2 from induction of anaesthesia until up to 5 min after intubation?
* A lower frequency of severe complications (severe arrhythmias, cardiac arrest, death)?
* A lower rate of intubation-related difficulties (change of method, change of operator, oesophageal intubation)?
* Decrease the duration of intubation (from laryngoscopy until end-tidal CO2 is registered)?
* Perceived difficulties, advantages and operator stress?

Design of study

This is and observational two-phase study, with the introduction of a checklist prior to phase two. The first phase will consist of a period of 6 to 8 months, and data regarding these intubations will be collected from the pre-existing quality register at the ICU. After this period, a checklist for intubation will be introduced and implemented, and endotracheal intubation will commence with the walkthrough of this cognitive aid. After the introduction of the checklist, the second phase of the study is started, where protocols on intubation will be collected and compared to the data from the first period.

Inclusion criteria

1. Adult, ≥18 years old
2. Intensive care patient that requires tracheal intubation for any indication

Exclusion criteria

1. Decided not suitable for any reason by the intensivist.
2. Under 18 years of age

If the checklist, for any reason, is not used for a patient after the implementation period, the data will still be included in the group of the second phase, since we believe the ICU staff will be considerably exposed to the checklist and hence, influenced by it.

Description of project This observational retrospective study will be conducted in the ICU, Karolinska University Hospital, Solna. The aim is to study whether introducing and implementing a pre-intubation checklist are associated with a lower incidence of intubation-related adverse events.

Adult ICU patients requiring intubation for any indication will be included, with inclusion and exclusion criteria as described above.

In a quality registry of ICU intubations, parameters such as pulse, blood pressure and SpO2 prior to, during and up to 5 minutes after intubation are manually registered from the monitor and put into the "ICU Respiration database". In addition, other intubation-related information is also registered, for instance: duration of intubation, airway assessment, intubation difficulty scale, intubation method and equipment, preoxygenation and intubation-related complications.

The study will consist of two phases. During the second phase, a checklist will be introduced and implemented based on the review of ICU airway guidelines and available literature. Physicians, residents and ICU nurses will receive information regarding the checklist prior to the intervention phase. If the checklist is not used for a patient during the second phase, the data will still be used in the cohort of the second group.

Data will be collected using the same intubation protocol as before the checklist introduction, containing patient demographics, the reason for ICU admission and intubation and vital parameters (saturation, blood pressure, pulse) before, during and after intubation. Blood gas analysis for arterial oxygen and carbon dioxide partial pressure will be analysed prior to intubation and in the immediate period after intubation (clinical practice). Furthermore, outcomes that will be registered are immediate complications such as desaturation, arterial hypotension, severe cardiac arrhythmia, cardiac arrest, death, oesophageal intubation, regurgitation, or a need for a surgical airway. Information regarding preoxygenation method, intubation circumstances and vasopressor use will be gathered, as well as 30-day mortality, length of hospital stay and ventilator days. Scores for physiological compromise ( and length of intensive care prior to intubation will be noted. Intubation-related data include the number of intubation attempts, Cormack-Lehane grade, time to end-tidal CO₂, the experience of the intubating physician, intubation difficulty scale, need for an alternative airway management and change of operator.

In both groups, the duration and method for preoxygenation and the drugs for anaesthetic induction are chosen as appropriate by the responsible intensivist.

Data will be collected from Clinisoft, the intensive care patient chart, regarding all intubations during the study period to find how many patients out of the total cohort that is not included during the study period.

The primary outcome is a comparison of intubation-related hypoxemic and hypotensive events between the two groups. Secondary events as severe arrhythmias, cardiac arrest, fatality and the number of intubation attempts will be analysed.

Statistics Data will be expressed as mean ± SD, median and range, 95% confidence intervals or number and percentage as appropriate. Comparison of two proportions will be performed using the chi-square test or Fischer exact test, where appropriate. Comparison of means will be performed using the student's t-test, while the comparison of medians will be analysed with the Mann-Whitney test. A p-value of <0.05 will be considered significant. Since this is a two-phase observational study of implementing a quality enhancing tool, it is, therefore, impossible to perform a correct power calculation. All the data, as mentioned above, will be compared between the two groups.

Clinical relevance Endotracheal intubation entails a significant risk of life-threatening complications in the intensive care setting. Therefore, optimising this procedure is of utmost importance. We aim to study whether the introducing and implementing a structured checklist for intubation will increase the safety of this standard yet perilous procedure. This could reduce the incidence of severe intubation-related complications and greatly benefit ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient in the ICU
* Need for tracheal intubation

Exclusion Criteria:

* Pateint is under 18 years of age
* Patiend inclusion is decided not suitable for any reason by the intensivist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive Care Patients that undergo tracheal intubation. All patients (before and after checklist) are registered with a protocol during intubation. This protocol is registered in a Respiratory Database.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Level of desaturation | From intubation up to 5 minutes after the procedure
  - Peripheral oxygen saturation (SpO2) below 90% (or >5% drop if saturation is <90% after preoxygenation).
Level of lowering blood pressure | From intubation up to 5 minutes after the procedure
  A systolic arterial pressure (SAP) below 90 mmHg

SECONDARY OUTCOMES:
30-day mortality | 30 days
Ventilator days | 30 days
  Amount of days on the ventilator in the intensive care unit
Days in the intensive care unit | 3 months
  A number describing the length of stay for the patient in the intensive care unit
Number of intubation attempts | 1 hour
  This describes how many attempts the anesthesiologist needs to complete intubation
First-pass success rate | 1 hour
  How many intubations succeed on the first try?
Lowest median oxygen saturation | From induction of anaesthesia until up to 5 min after intubation?
  Lowest median oxygen saturation after intubation
Number of arrythmias | Up to 5 min after intubation
  Asystole, bradycardia, takyarrythmia
Presence of cardiac arrest | Up to 5 minutes after intubation
  Circulatory arrest
Change of intubation method | 1 hour
  Does the method of intubation (laryngoscopy with tube, laryngeal device, thracheostomy) need to be abandoned or changed?
Change of operator during intubation? | During intubation
  New operator due to failure of the first one?
Intubation time | 5 minutes
  Time from laryngoscopy until end-tidal CO2 is registered

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Perioperative Medicine and Intensive Care, Stockholm, Sweden

REFERENCES:
- [Derived] Nejatian A, Forsberg IM, Thoro U, Sjoblom A, Kahlin J. Impact of Checklist Implementation on Endotracheal Intubation-Related Complications in Critically Ill Adults-A Retrospective Before and After Study. Acta Anaesthesiol Scand. 2025 Aug;69(7):e70103. doi: 10.1111/aas.70103. PMID 40692385